CLINICAL TRIAL: NCT02693067
Title: A Phase 1 Study to Assess the Safety, Tolerability and Effectiveness of PV-10 Chemoablation of Neuroendocrine Tumours (NET) Metastatic to the Liver in the Reduction of Biochemical Markers and Symptoms Caused by Secretory Products
Brief Title: A Phase 1 Study of PV-10 Chemoablation of Neuroendocrine Tumours (NET) Metastatic to the Liver
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Provectus Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Provectus Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PV-10-NET-01
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Neuroendocrine Tumors Metastatic to the Liver
MeSH Terms: interventions — Rose Bengal B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PV-10 (Experimental): Intralesional rose bengal disodium (PV-10) to one or more neuroendocrine tumor metastases to the liver
  Interventions: Drug: Rose bengal disodium

INTERVENTIONS:
Drug: Rose bengal disodium — Percutaneous intralesional injection to NET tumor
  Other Names: PV-10

SUMMARY:
This study is intended to determine the safety, tolerability and reduction of biochemical markers (Chromogranin A or, if deemed appropriate, 5-hydroxyindoleaceticacid) and troublesome symptoms (particularly diarrhea and flushing) of intralesional injection of PV-10 in subjects with NET metastatic to the liver that are not amenable to resection or other potentially curative therapy.

DETAILED DESCRIPTION:
This is a single center, open-label study to evaluate the safety, tolerability, and effect on tumor growth and symptomology (clinical and biomarkers) following a single intralesional injection of PV-10 in subjects with neuroendocrine tumors metastatic to the liver. Subjects will be divided into two cohorts (up to 6 subjects in each), the first of which will receive intralesional PV-10 to one liver lesion (to a maximum dose of 15 mL PV-10) to assess safety. If safety is established, cohort two will receive treatment to all amenable lesions (to a maximum dose of 15 mL PV-10). Subjects can have further lesions treated 6 weeks after their initial treatment provided any preceding treatments with PV-10 were well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, males and females.
2. Histologically or cytologically confirmed, or clinically diagnosed based on currently accepted standards, NET tumors metastatic to the liver that are not amenable at the time of enrolment to resection, transplant or other potentially curative therapy. Patients must have at least one common NET symptom (European Organization for Research and Treatment of Cancer GI.NET21 instrument score of 2 or more at baseline) including: flushing, diaphoresis, diarrhea, abdominal discomfort, hyperacidity, dyspnea or palpitations.
3. The Target Lesion(s) must be determined to be amenable to percutaneous injection by the treating physician.
4. The Target Lesion(s) must have measurable disease, defined as a unidimensionally measurable lesion ≥ 1.0 cm in longest diameter by helical computed tomography (CT); the maximum diameter of any Target Lesion should be ≤ 3.9 cm. These lesions should also overexpress SSTR. If the lesion is negative on positron emission tomography-computed tomography (PET/CT), there is no need to perform further PET/CT scans.
5. Performance status of Karnofsky scale 60%-100% or Eastern Cooperative Oncology Group (ECOG) performance scale 0-2.
6. Life expectancy ≥ 6 Months.
7. Hematopoietic Function

   * White blood cells (WBC) ≥ 2,500/mm3.
   * Absolute neutrophil count (ANC) ≥ 1000/mm3.
   * Hemoglobin ≥ 8 g/dL.
   * Platelet count ≥ 50,000/mm3.
   * Coagulation: international normalized ratio (INR) ≤ 1.3.
8. Blood Chemistry

   * Aspartate transaminase (AST) and alanine transaminase (ALT) < 5 times Upper Limit of Normal (ULN).
   * Alkaline phosphatase (ALP) < 5 times ULN.
   * Bilirubin ≤ 1.5 times ULN.
   * Creatinine ≤ 1.5 times ULN and estimated glomerular filtration rate (eGFR) ≥ 50.
9. Thyroid Function

   • Total T3 or free T3 (serum triiodothyronine), total T4 or free T4 (serum thyroxine) and TSH (serum thyrotropin) ≤ Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 abnormality.
10. Renal Function

    • Subjects must have adequate renal function in the opinion of the Investigator with no clinically significant renal impairment or uncontrolled renal disease, see 8 above.
11. Cardiovascular Function

    • Subjects must have adequate cardiovascular function in the opinion of the Investigator with no clinically significant uncontrolled cardiovascular disease. All subjects must have a cardiac echo performed within 12 months to exclude tricuspid incompetence ("carcinoid heart syndrome").
12. Respiratory Function

    • Subjects must have adequate respiratory function in the opinion of the Investigator with no clinically significant uncontrolled respiratory disease.
13. Immunological Function

    • Subjects must have adequate immune system function in the opinion of the Investigator with no known immunodeficiency disease.
14. Long Acting Somatostatin Analogs

    • Subjects on long acting somatostatin analogs must be stable on treatment. Somatostatin analogs are to be continued throughout the study period.
15. Informed Consent: Signed by the subject prior to screening.

Exclusion Criteria:

1. Target Lesion(s) must not be contiguous with, encompass or infiltrate major blood vessels.
2. Liver metastases amenable to resection, transplant or other potentially curative therapy.
3. Subjects who have received hepatic surgery, ablation or chemoembolization within 4 weeks of PV-10 administration.
4. Radiation Therapy • Subjects who have received hepatic radiation within 4 weeks of PV-10 administration.
5. Chemotherapy

   • Subjects who have received chemotherapy within 4 weeks of PV-10 administration (6 weeks for nitrosoureas or mitomycin C).
6. Investigational Agents

   • Subjects who have received investigational agents within 4 weeks (or 5 half-lives) of PV-10 administration.
7. Phototoxic or Photosensitizing Agents

   • Subjects who have received agents posing a clinically significant risk of photosensitivity reaction within 5 half-lives of PV-10 administration.
8. Concurrent or Intercurrent Illness

   * Subjects with significant concurrent or intercurrent illness, psychiatric disorders or alcohol or chemical dependence that would, in the opinion of the Investigator, compromise their safety or compliance or interfere with interpretation of the study.
   * Subjects with uncontrolled thyroid disease or cystic fibrosis.
   * Presence of clinically significant acute or unstable cardiovascular, cerebrovascular (stroke), renal, gastrointestinal, pulmonary, immunological (with the exception of the presence of hepatitis B virus (HBV), viral hepatitis, or cirrhosis), endocrine, or central nervous system disorders.
   * Current encephalopathy or current treatment for encephalopathy.
   * A documented variceal hemorrhage within 4 months of screening.
   * History of human immunodeficiency virus or acquired immune deficiency syndrome.
   * The clinical or radiological presence of ascites.
9. Pregnancy

   * Female subjects who are pregnant or lactating.
   * Female subjects who have positive serum pregnancy test taken within 7 days of PV-10 administration.
   * Fertile subjects who are not using effective contraception (e.g., oral contraceptives, intrauterine devices, double barrier methods such as condoms and diaphragms, abstinence or equivalent measures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2021-09-01 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 28 days
  Incidence of Systemic and Locoregional Adverse Events will be Coded and Tabulated

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  Response of Injected Target and Measurable Bystander Lesions (if present) will be Tabulated
Target Lesion Somatostatin Receptor (SSTR) Expression | 6 months
  Change in SSTR Expression will be Assessed vs Baseline Values
Change in Neuroendocrine Tumor Biomarkers | 6 months
  Change in Chromogranin A (CgA) and/or 5-Hydroxyindole Acetic Acid (5-HIAA) will be Assessed vs Baseline Values
Reduction in Major Symptoms | 6 months
  Change in Major Symptoms (Diarrhea and Flushing) will be Separately Assessed using European Organization for Research and Treatment of Cancer QLQ-C30 and GI.NET21 Symptom Scores vs Baseline Values
Reduction in Other Symptoms | 6 months
  Change in Other Symptoms (including Bronchoconstriction and Abdominal Cramping) will be Separately Assessed using QLQ-C30 and GI.NET21 Symptom Scores vs Baseline Values
Change in Peripheral Blood Mononuclear Cells (PBMC) | 28 days
  Change in PBMC will be Assessed vs Baseline Values

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wachter, Ph.D., Study Director — Provectus Biopharmaceuticals, Inc.
Locations (1):
- The Queen Elizabeth Hospital, Woodville, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Price T, Depauw L, Cehic G, Wachter E, Sebben R, Reid J, Neuhaus S, Alawawdeh A, Kirkwood ID, Solanki R, McGregor M, Leopardi L, Rodrigues D, Maddern G. A phase 1 study to assess the safety, tolerability and effectiveness of PV-10 (Rose Bengal Sodium) in neuroendocrine tumours metastatic to the liver. Br J Cancer. 2025 Jun;132(10):888-896. doi: 10.1038/s41416-025-02976-9. Epub 2025 Mar 26. PMID 40140696